CLINICAL TRIAL: NCT04460469
Title: Self-assessment of Anxiety Level and Oral Hygiene Practice in Dental Students of Cairo University During Covid-19 Pandemic
Brief Title: Anxiety Level and Oral Hygiene Practice in Dental Students During Covid-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Zakaria Ibrahium Mohammed, Lecturer Oral Medicine & Periodontology, Faculty of Dentistry, Cairo University, Cairo University
Other Study IDs: Mai Zakaria 4
Record Dates: First submitted 2020-07-04; First posted 2020-07-07 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Anxiety; Covid19; Oral Hygiene
Keywords: Anxiety; Covid19; Oral Hygiene Practice; Dental students; questionnaire
MeSH Terms: conditions — Anxiety Disorders; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Covid-19, the infection caused by a novel corona virus detected in December 2019 in Wuhan (Hubei province), is now a pandemic announced by World Health Organization, raising concerns of widespread panic and increasing anxiety in individuals. This outbreak results in mass quarantine in Egypt since middle of March 2020. Brooks et al. (2019) reviewed and reported quarantine could bring "post traumatic stress symptoms, confusion, and anger. Stressors included longer quarantine duration, infection fears, frustration, boredom, inadequate supplies, inadequate information, financial loss, and stigma.". Many universities decided to suspend in-person classes and evacuate students in responding to the intensifying concerns surrounding Covid-19. This action can lead to negative psychological consequences among college students. Oral health related behavior and attitudes habits correlate with oral health status and can be considered to be its predictors . There is a claim of potential connection between high bacterial load in the mouth and complications associated with Covid-19 infection. Bacteria present in the meta genome of patients severely infected with Covid-19 included high reads for Prevotella, Staphylococcus, and Fusobacterium, all usually commensal organisms of the mouth. Over 80% of patients in ICU exhibited an exceptionally high bacterial load. Accordingly, the investigators assume that good oral hygiene better to be maintained during a Covid-19 outbreak in order to reduce the bacterial load in the mouth and the risk of a bacterial super infection in case of catching the infection .

While there seems to be a common belief that psychosocial stress affects oral hygiene behavior, this assumption has rarely been proved9 Dental students, as the future providers of dental care, are ex¬pected to be role models for their patients regarding the oral hygiene practice and they supposed to be aware of the importance of preserving the oral health. Thus, we intended to select them as our population to study how the level of anxiety during pandemic could affect the practice of oral hygien

DETAILED DESCRIPTION:
A cross sectional study (survey) will be conducted among dental students in faculty of dentistry Cairo University for the duration of one month from June 2020 to July 2020.

The questionnaire has three parts. The first part included demographic details. The second part included validated general anxiety disorder scale GAD-7. Questionnaire consisting of seven questions which measures students' anxiety level score. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. The third part the validated self administered, structured, and close ended 15 questions that assessed the self reported oral hygiene practices 11. The questionnaire forms were kept anonymous. The questionnaire was validated.

ELIGIBILITY:
Inclusion Criteria:

* Student of faculty of Dentistry, Cairo University

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The questionnaire is going to be disseminated as google form to all the Cairo university dental students via emails .
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
correlate between the level of anxiety and the practice of oral hygiene during covid-19 pandemic in dental students of Cairo university | 2 months
  By questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mai Zakaria, Ph, Principal Investigator — Lecturer Oral Medicine & Periodontology, Faculty of Dentistry, Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
individual participant data are not to be shared with other researchers until publication of the study.